CLINICAL TRIAL: NCT03560778
Title: Comparisons of Urodynamic, Bladder Diary, Quality of Life Parameters Between OAB-wet and OAB-dry Female Patients
Acronym: OAB
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201404012RINC
Record Dates: First submitted 2018-04-25; First posted 2018-06-18 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-04

CONDITIONS: Urinary Bladder, Overactive
Keywords: Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urodynamics
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A small bladder capacity and more frequent urgency episodes were predictors of OAB-wet, and the above findings might indicate that OAB-wet and OAB-dry are a continuum of OAB. Older age, high maximum flow rate, high detrusor pressure at maximum flow rate and the presence of urodynamic stress incontinence were also independent predictors for OAB-wet, and the above might indicate that OAB-wet and OAB-dry have at least partly different underlying pathophysiologies.

DETAILED DESCRIPTION:
Aims: To identify factors predicting the presence of OAB-wet and to further derive the underlying pathophysiology in OAB-wet vs. OAB-dry.

Methods: Between September 2007 and September 2013, the medical records of women with OAB who completed a 3-day bladder diary and underwent urodynamic studies in a tertiary referral center will be reviewed. OAB-wet will be diagnosed in patients who complained of at least one episode of urgency incontinence in the previous month; otherwise, OAB-dry is diagnosed. Multivariate logistic regression analysis will be used to predict the presence of OAB-wet.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of overactive bladder disease
2. Female patient of more than 20 year-old

Exclusion Criteria:

1. Dominant symptoms with stress urinary incontinence (SUI)
2. Regular urethral catheterization or intermittent self-catheterization
3. Urinary tract infection or chronic inflammation in the previous 2 weeks
4. Bladder calculus
5. A history of pelvic radiotherapy
6. A preexisting malignant pelvic tumor.

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with OAB who completed a 3-day bladder diary and underwent urodynamic studies at the urogynecologic outpatient clinics of the Department of Obstetrics and Gynecology of a medical center
Sampling Method: Non-Probability Sample
Enrollment: 623 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Compare the difference of urodynamic parameters between OAB-wet and OAB-dry | 1 week
  The variables of urodynamic study included maximum flow rate, average flow rate, voided volume, volume of strong to desire, detrusor pressure at maximum flow during voiding cystometry (PdetQmax), Valsalva leak point pressure (VLPP), maximal urethral pressure (MUP), maximal urethral closure pressure (MUCP), functional profile length, urethral closure pressure area (UCPA), continence length, continence area, pressure transmission ratio (PTR) at MUP, and electromyography (EMG). The urodynamic parameters will be interpreted together to get a complete urodynamic report and diagnosis, thus to compare the difference between OAB-wet and OAB-dry
Compare the difference of bladder diary parameters between OAB-wet and OAB-dry | 1 week
  The 3-day bladder diary parameters included maximum daytime voided volume excluding the morning void derived from 3-day bladder diaries (DVVmax), urgency episodes, urgency incontinence episodes, daytime frequency, nocturia, total voided volume and total water intake. The bladder diary parameters will be interpreted together to get a complete report, such as urinary urgency and nocturia, thus to compare the difference between OAB-wet and OAB-dry